CLINICAL TRIAL: NCT06679192
Title: Comparing a Thickness-Varied Soft Surface of Custom Made Shoe Insoles Based on Plantar Pressure Analysis in Shoes, to Insoles With Even Thickness Surfaces: A Cross Sectional Study Design
Brief Title: Thickness-Varied Soft Surface on Shoe-Insoles Based on In-Shoe Pressure Measurement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2024-02115-01
Record Dates: First submitted 2024-11-04; First posted 2024-11-07 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-11

CONDITIONS: Diabetes Mellitus
Keywords: plantar pressure; shoe insert; ulcer prevention
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: three-intervention cross over study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Thickness-Varied soft surface insole (Experimental): Each participant will be measured with this insole. The order between the three insoles is randomized.
  Interventions: Device: Milled thickness varied soft upper surface, based on plantar pressure measurement
- 3mm soft surface insole (Experimental): Each participant will be measured with this insole. The order between the three insoles is randomized.
  Interventions: Device: 3mm soft upper surface
- No soft surface insole (Experimental): Each participant will be measured with this insole. The order between the three insoles is randomized.
  Interventions: Device: No soft upper surface

INTERVENTIONS:
Device: Milled thickness varied soft upper surface, based on plantar pressure measurement — This custom made shoe insole is milled, with a thickness varied soft upper surface ranging from 0-6mm in thickness. The base of the insole is 45 shore Ethylene-vinyl acetate (EVA).
  This intervention makes the insole from an individual foot scan, a plantar pressure measurement from the individual and the shoe model to mill a finished custom made shoe insole with a soft upper surface. It is difficult in clinical practice of making shoe inserts to create a thickness varied soft upper with different zones all over the insole. Furthermore, a soft upper requires a physical positive model to be made of the foot and staff must spend time to grind the insole to an acceptable shape. A milled version would be more effective since it require no physical foot model, little to no work grinding the insole and enables the use of thickness-variations. It also enables the use of data-based insole-manufacturing, such as data from plantar pressure measurements.
  Arms: Thickness-Varied soft surface insole
Device: 3mm soft upper surface — This intervention has a 3mm soft layer on the insole, milled with a 45 shore base of the custom made insole. This is one of the most commonly used designs in clinical practice.
  Arms: 3mm soft surface insole
Device: No soft upper surface — This intervention has a no soft layer on the insole, milled with a 45 shore base of the custom made insole. This is one of the most commonly used designs in clinical practice.
  Arms: No soft surface insole

SUMMARY:
The goal of this cross-sectional study is to evaluate a new shoe insole manufacturing method with the goal of further preventing foot ulceration for people with diabetes. This is achieved by decreasing pressure under risk areas of the foot, often on the insole; the interface between the shoe and the foot. The main question it aims to answer is:

Does a thickness-varied surface based on plantar pressure measurement decrease pressure at high risk areas compared to even thickness surfaces.

Researchers will compare three different pairs of insoles for each participant.

Participants will partake in two sessions. The first one being a pre-measurement and foot status for manufacturing the insoles. During the second session, three pairs of insoles will in a random order be tested for each participant. The pressure measurement of the insoles will be made using F-Scan(TM), while participants walk.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age at the date of signing consent.
* Diabetes mellitus 1 or 2
* Diabetic foot risk group 2: Signs of distal neuropathy and/or peripheral circulatory disorder.
* Able to walk 10 meters without walking aids
* Able to speak and understand Swedish

Exclusion Criteria:

* Diabetic foot risk group 3: Distal neuropathy or peripheral circulatory disorder and foot ulcers, or amputation, foot deformity of clinical importance or skin pathology.
* Diabetic foot risk group 4: Occuring foot ulcer, severe osteoarthropathy or chronic foot pain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-11-11 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Plantar pressure | Pre-measurement used for insole design at first meeting. Intervention-measurement for all patients and interventions at second meeting, approximately 3-4 weeks after pre-measurement.
  Measured plantar pressure (kPa) differences between the arms/interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Roy Tranberg, PhD, Docent, Principal Investigator — Vastra Gotaland Region
Locations (1):
- TeamOlmed Hagaplan, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No